CLINICAL TRIAL: NCT04515251
Title: A Prospective, Observational, Multicenter Study on Ultrasound Evaluation of Superior Mesenteric Artery Measurements in a Healthy Pediatric Population
Brief Title: Ultrasound Evaluation of Superior Mesenteric Artery Measurements in a Healthy Pediatric Population
Status: Recruiting | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Collaborators: Imaging Institute of Southern Switzerland (Unknown)
Responsible Party: Principal Investigator, Marirosa Cristallo Lacalamita, MD Principal investigator, Ente Ospedaliero Cantonale, Bellinzona
Other Study IDs: RAD-SMA-001
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Superior Mesenteric Artery Syndrome
MeSH Terms: conditions — Superior Mesenteric Artery Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Ultrasound measurements — ultrasound measurement at the level of the left renal vein on a sagittal plane according to age

SUMMARY:
Multicenter, prospective, observational research project on children aged from 10 to 15 years old undergoing abdominal ultrasound examinations during routine clinical practice.

DETAILED DESCRIPTION:
Demographics data, clinical indications, ultrasound diagnosis, and ultrasound measurements will be recorded and stored on an database. Ultrasound measurements will be analyzed to define the normal range of values of Superior Mesenteric Artery (SMA) angle and Superior Mesenteric Artery - Aorta (SMA-A) distance in the pediatric population according to age, Body Mass Index (BMI), and fat parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children
* Age ranging from10 to 15 years, included
* Abdominal ultrasound examination to be performed for indications other than gastrointestinal evaluation
* Signed Informed Consent

Exclusion Criteria:

* Presence of a disease that could distort the anatomy around the SMA (e.g., abdominal mass, lymphadenopathy, severe scoliosis, free abdominal fluid)
* Oncologic patients at risk of neoplastic cachexia.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged from 10 to 15 years
Sampling Method: Non-Probability Sample
Enrollment: 289 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Define the normal range of values of the SMA angle | 1 day
  Measurement in degree with its 95% confidence interval

SECONDARY OUTCOMES:
Define the normal range of values of the SMA-A distance LV | 1 day
  Measurement in millimeter (mm) with its 95% confidence interval measured through ultrasound examination at the level of the left renal vein on an axial plane according to age
Define the normal range of values of the SMA-A distance D | 1 day
  Measurement in millimeter (mm) with its 95% confidence interval measured through ultrasound examination at a level where the third part of the duodenum crosses on an axial plane according to age
Define the normal range of values of the SMA angle (degree), SMA-A distance LV | 1 day
  Measurement in millimeter (mm) with its 95% confidence interval measured through ultrasound examination according to BMI categories, subcutaneous and visceral fat thickness
Assess the association between the SMA angle and BMI categories | 1 day
  According to age and sex.

CONTACTS AND LOCATIONS:
Overall Officials: Marirosa Cristallo Lacalamita, MD, Principal Investigator — Imaging Institute of Southern Switzerland
Locations (2):
- Switzerland (2):
  - Imaging Institute of Southern Switzerland, Bellinzona
  - Hôpitaux Universitaires Genève, Geneva

IPD SHARING:
Plan to Share IPD: No